CLINICAL TRIAL: NCT02213458
Title: University of California, San Francisco (UCSF) and University of Nebraska Medical Center (UNMC) Care Ecosystem
Brief Title: Care Ecosystem: Navigating Patients and Families Through Stages of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Nebraska (Other); Centers for Medicare and Medicaid Services (U.S. Federal Agency); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1C12013003302; 5R01AG056715 (NIH); 1C1CMS331346 (Other Grant/Funding Number: Centers for Medicare and Medicaid Services)
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Dementia; Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Frontotemporal Lobar Degeneration; Memory Disorders
Keywords: Pragmatic Clinical Trial; Family Caregivers; Patient Care Management
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Frontotemporal Lobar Degeneration; Memory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Navigated Care (Experimental): Comprehensive longitudinal continuing care program
  Interventions: Behavioral: Navigated Care
- Survey of Care (No Intervention): Control group that will undergo the same regular assessments as patients enrolled in Navigated Care

INTERVENTIONS:
Behavioral: Navigated Care — Navigated Care emphasizes continuous and personalized care and is based on 3 modules: the Caregiver Module that includes educational interventions and connects families with community resources, the Decision-Making Module that facilitates proactive medical, financial, and safety decisions, and the Medication Module that identifies inappropriate medication usage via pharmacist review. Innovative technology in the form of a "dashboard" functions as a patient care management system used by Care Team Navigators (CTNs).
  Arms: Navigated Care

SUMMARY:
This is a randomized clinical trial evaluating the benefits of a program that supports model care for persons with dementia and their family caregivers. Subjects were recruited from California, Nebraska and Iowa. Subjects determined to be eligible were consented and randomized into one of two groups. Two thirds of patients were enrolled into Navigated Care that provided them with assistance in meeting important benchmarks in their care, for example completion of legal and financial planning and strategies for minimizing caregiver burden. One third of patients were enrolled to a control group, entitled Survey of Care. Outcomes include quality of life, health care utilization, caregiver burden, satisfaction with care, caregiver depression, and caregiver self-efficacy.

ELIGIBILITY:
This study will enroll patients as well as their primary caregivers as research participants.

Inclusion criteria for patient participants:

1. Patient has a diagnosis of dementia with a progressive course
2. Patient has a primary caregiver (identified as having primary responsibility for patient) that is eligible for and agrees to join the study
3. Patient is covered by Medicare or Medi-caid or is Medi-pending
4. Patient is expected to live at least 3 months based on assessment by the referring provider, the patient's primary care provider, or medical record review
5. Patient speaks either English, Cantonese, Mandarin, or Spanish
6. Patient lives in California or Nebraska or Iowa
7. Patient is age 45 or older

Inclusion criteria for caregiver participants:

1. Caregiver has primary responsibility for dementia patient that is eligible for and agrees to join the study
2. Caregiver speaks either English, Cantonese, Mandarin, or Spanish
3. Caregiver is a legal adult

Exclusion Criteria:

1. Patient resides in a nursing home or skilled nursing facility at time of enrollment
2. Participant is enrolled in a similar clinical trial that precludes their participation in our trial
3. Patient is pregnant

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Possin, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Nebraska Medical Center, Omaha, Nebraska

REFERENCES:
- [Result] Guterman EL, Kiekhofer RE, Wood AJ, Allen IE, Kahn JG, Dulaney S, Merrilees JJ, Lee K, Chiong W, Bonasera SJ, Braley TL, Hunt LJ, Harrison KL, Miller BL, Possin KL. Care Ecosystem Collaborative Model and Health Care Costs in Medicare Beneficiaries With Dementia: A Secondary Analysis of a Randomized Clinical Trial. JAMA Intern Med. 2023 Nov 1;183(11):1222-1228. doi: 10.1001/jamainternmed.2023.4764. PMID 37721734
- [Result] Liu AK, Possin KL, Cook KM, Lynch S, Dulaney S, Merrilees JJ, Braley T, Kiekhofer RE, Bonasera SJ, Allen IE, Chiong W, Clark AM, Feuer J, Ewalt J, Guterman EL, Gearhart R, Miller BL, Lee KP. Effect of collaborative dementia care on potentially inappropriate medication use: Outcomes from the Care Ecosystem randomized clinical trial. Alzheimers Dement. 2023 May;19(5):1865-1875. doi: 10.1002/alz.12808. Epub 2022 Nov 4. PMID 36331050
- [Result] Possin KL, Merrilees JJ, Dulaney S, Bonasera SJ, Chiong W, Lee K, Hooper SM, Allen IE, Braley T, Bernstein A, Rosa TD, Harrison K, Begert-Hellings H, Kornak J, Kahn JG, Naasan G, Lanata S, Clark AM, Chodos A, Gearhart R, Ritchie C, Miller BL. Effect of Collaborative Dementia Care via Telephone and Internet on Quality of Life, Caregiver Well-being, and Health Care Use: The Care Ecosystem Randomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1658-1667. doi: 10.1001/jamainternmed.2019.4101. PMID 31566651

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Navigated Care | Survey of Care
Started | 1024 | 536
Completed | 970 | 526
Not Completed | 54 | 10
Not completed — No longer meets criteria: caregiver deceased | 4 | 0
Not completed — No longer meets criteria: caregiver no longer caregiving | 4 | 0
Not completed — No longer meets criteria: caregiver too sick to participate | 2 | 0
Not completed — No longer meets criteria: patient moved out of state | 10 | 0
Not completed — Refused re-consent | 6 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 26 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Navigated Care | Survey of Care | Total
Number analyzed (Participants) | 1024 | 536 | 1560
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 241 | 157 | 398
  >=65 years | 783 | 379 | 1162
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.1 (8.66) | 78.1 (12.0) | 78.1 (9.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 656 | 336 | 992
  Male | 226 | 200 | 426
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 107 | 58 | 165
  Not Hispanic or Latino | 911 | 477 | 1388
  Unknown or Not Reported | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 73 | 29 | 102
  Native Hawaiian or Other Pacific Islander | 5 | 1 | 6
  Black or African American | 45 | 19 | 64
  White | 825 | 447 | 1272
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 72 | 37 | 109
Region of Enrollment [Number; unit: participants]
  United States | 1024 | 536 | 1560

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life-Alzheimer's Disease, Change From Baseline to 1 Year
Description: An established 13-item measure, with a 1-4 ordinal scale for each item, to obtain a rating of the patient's quality of life from the caregiver. Item scores are summed for a total score ranging from 13-52, with higher scores representing better quality of life
Time Frame: Baseline to one year
Population: The subset of caregivers with completed QDRS and Quality of Life questionnaires at baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Navigated Care | Survey of Care
Number analyzed (Participants) | 504 | 261
units on a scale | -1.43 (5.64) | -1.12 (5.87)
Statistical Analysis 1: Comparison: Navigated Care vs Survey of Care; Linear mixed effects model; Test type: Superiority; p = 0.04, Mixed Models Analysis; Controlling for dementia severity (QDRS); Slope = .539, 95% CI 2-sided [.259 to 1.337]

2. Secondary Outcome: Change in Caregiver Reported Rate of Emergency Department Utilization: Baseline to One Year
Description: Health care utilization based upon caregiver survey to assess emergency department, hospitalization, and ambulance use rates. To be confirmed using Medicare claims data.
Time Frame: Baseline to one year
Population: Subset of patients with complete data on QDRS and emergency department visits at baseline
Measure: Mean (Standard Deviation); unit: number of encounters
Arm/Group | Navigated Care | Survey of Care
Number analyzed (Participants) | 503 | 261
number of encounters | .0483 (.703) | .175 (.840)
Statistical Analysis 1: Comparison: Navigated Care vs Survey of Care; Test type: Superiority; p = .05, Mixed Models Analysis; Linear mixed model controlling for dementia severity (QDRS); Slope = -.138, 95% CI 2-sided [-.295 to -.020]

3. Secondary Outcome: Change in Caregiver Burden, Baseline to One Year
Description: Zarit Burden Interview (short version). An established 12-item measure, with a 0-4 ordinal scale for each item, to measure caregiver burden. Item scores are summed for a total score ranging from 0-48, with higher scores representing higher levels of burden.
Time Frame: Baseline to one year
Population: Subset of patients with complete data on QDRS and Zarit burden at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Navigated Care | Survey of Care
Number analyzed (Participants) | 503 | 262
score on a scale | -1.682 (8.144) | -1.482 (8.641)
Statistical Analysis 1: Comparison: Navigated Care vs Survey of Care; Test type: Superiority; p = 0.07, Mixed Models Analysis; Linear mixed model controlling for dementia severity (QDRS); Slope = -1.902, 95% CI 2-sided [-3.885 to -0.080]

4. Secondary Outcome: Satisfaction With Dementia Care
Description: A novel 1-item measure, with a 1-5 ordinal scale, to measure caregiver satisfaction with dementia care provided by the patient's clinical team. Also, one question asking caregivers whether they would recommend the Care Ecosystem to another caregiver. Collected in the treatment group only.
Time Frame: One year
Population: Navigated Care caregivers with completed caregiver satisfaction questionnaire at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Navigated Care
Number analyzed (Participants) | 325
Participants
  Very satisfied with Care Ecosystem services | 148
  Satisfied with Care Ecosystem services | 107
  Neutral toward Care Ecosystem services | 57
  Unsatisfied with Care Ecosystem services | 9
  Very unsatisfied with Care Ecosystem services | 4

5. Secondary Outcome: Change in Caregiver Depression, Baseline to One Year
Description: Patient Health Questionnaire 9 (PHQ-9). Higher scores represent more severe depression. Scores range from 0-27.
Time Frame: Baseline to one year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Navigated Care | Survey of Care
Number analyzed (Participants) | 503 | 262
score on a scale | -0.831 (4.312) | -0.238 (4.053)
Statistical Analysis 1: Comparison: Navigated Care vs Survey of Care; Test type: Superiority; p = 0.03, Mixed Models Analysis; Slope = -1.143, 95% CI 2-sided [-2.154 to -0.132]

6. Secondary Outcome: Change in Caregiver Self-efficacy, Baseline to One Year
Description: A novel 4-item measure on a 1-5 ordinal scale to measure self-efficacy around dementia caregiving. Higher scores represent greater self-efficacy. Scores range from 5-15.
Time Frame: Baseline to one year
Population: Dyads with baseline data on dementia severity (QDRS) and self-efficacy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Navigated Care | Survey of Care
Number analyzed (Participants) | 503 | 262
units on a scale | 1.356 (3.038) | 1.043 (2.647)
Statistical Analysis 1: Comparison: Navigated Care vs Survey of Care; Test type: Superiority; p = 0.11, Mixed Models Analysis; Controlling for dementia severity (QDRS); Slope = .635, 95% CI 2-sided [-0.135 to 1.405]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Navigated Care | Survey of Care
All-Cause Mortality (participants affected / at risk) | 74/1024 | 39/536
Serious Adverse Events (participants affected / at risk) | 269/1024 | 143/536
Other Adverse Events (participants affected / at risk) | 0/1024 | 0/536
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navigated Care (N=1024) | Survey of Care (N=536)
Overnight hospitalization (General disorders) | 218 (433) | 116 (194)
Severe fall (General disorders) | 51 (57) | 32 (34) — Falls resulting in major injury (broken bone, major bleeding, or loss of consciousness)

LIMITATIONS AND CAVEATS:
The economic outcomes are not reported beyond 12-month follow-up and were based only on survey data. Our sample likely differs in important ways from samples from similar programs that do not have a randomized control condition. During our recruitment and consent process, the only potential benefit communicated to prospective enrollees was that participation might inform and advance the quality of care provided to patients with dementia (PWDs) and their caregivers in the future.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT02213458/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT02213458/SAP_001.pdf